CLINICAL TRIAL: NCT00105495
Title: Randomized Trial Comparing the Relative Efficacy of Deferiprone to That of Deferoxamine in Removing Excess Cardiac Iron in Thalassemia Major Patients
Brief Title: Efficacy Study in Removing Excess Iron From the Heart
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ApoPharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LA16-0102
Record Dates: First submitted 2005-03-15; First posted 2005-03-16 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2006-10

CONDITIONS: Thalassemia Major; Hemosiderosis
Keywords: Iron Overload; Thalassemia; Haemosiderosis; Cardiac; Deferiprone; Chelation
MeSH Terms: conditions — beta-Thalassemia; Hemosiderosis; Iron Overload; Thalassemia; Hemochromatosis | interventions — Deferiprone; Deferoxamine

INTERVENTIONS:
Drug: Ferriprox (deferiprone)
Drug: Desferal (deferoxamine)

SUMMARY:
The purpose of this study is to determine whether deferiprone has superior efficacy in removing excess iron from the heart when compared with deferoxamine.

DETAILED DESCRIPTION:
This study is a multi-center, randomized, open-label, controlled clinical trial. The study population is participants with thalassemia major who are receiving regular chelation therapy with deferoxamine. A total of sixty (60) participants will be enrolled among the investigative sites.

The primary objective of this study is to determine whether deferiprone exhibits superior efficacy in removing excess iron from the heart compared to that of the standard therapy, deferoxamine.

The secondary objective is to evaluate the relative efficacy of deferiprone with respect to that of deferoxamine as assessed by serum ferritin concentration and liver iron concentration.

The primary efficacy measure in this study will be the participants' cardiac iron status, as determined by heart MRI T2* assessments.

The secondary efficacy measure will be by serum ferritin concentration and liver iron concentration. This will be measured by the Superconducting Quantum-Interference Device (SQUID) BioSusceptometer.

The duration of treatment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of thalassemia major as confirmed by laboratory and clinical criteria
* Participants who are well transfused-maintaining a mean pre-transfusion Hb (hemoglobin) no less than 9 g/dL.
* Between 18 and 36 years of age.
* Receiving ongoing chelation therapy with deferoxamine for at least the past five years. Those who have been exposed to deferiprone for

  ≤ 6 months but not within the last 2 years prior to commencement of this study will be considered eligible to participate.
* Abnormal heart MRI T2* greater than or equal to 8 ms and < 20 ms.
* If female, fertile, and is neither pregnant nor lactating, confirms she will use an effective method of contraception for the length of the trial and has a negative pregnancy test immediately prior to commencement of study drug OR has had a tubal ligation OR a hysterectomy OR is post menopausal (at least 1 year no menses prior to enrollment in the study) OR their only sexual partner has been sterilized (if male).
* If male and fertile, he confirms that he and/or his partner will use an effective method of contraception for the length of the trial.
* Provide a signed and witnessed written informed consent obtained prior to the first study intervention.

Exclusion Criteria:

* Have anemia other than thalassemia.
* HIV antibody positive.
* Clinical evidence of cardiomyopathy as shown by LV Shortening Fraction < 30 % and/or CMR derived LV (left ventricular) Ejection Fraction < 56 %.
* Severe/significant arrhythmia, including those who have had atrial fibrillation (participants with occasional ectopic beats and normal echo can be included) or those requiring treatment.
* Previously discontinued therapy with deferiprone or deferoxamine because of an adverse drug reaction to either chelator.
* Have received deferiprone in the last five years. However those who have been exposed to deferiprone for ≤ 6 months but not within the last 2 years prior to commencement of this study will be considered eligible to participate.
* Evidence of abnormal liver function (liver enzymes > 3 times upper limit of normal - entry may be delayed until return to normal).
* Have disorders associated with neutropenia (ANC < 1.5 x 10^9/L) or thrombocytopenia (platelet count <50 x 10^9/L) in the twelve months prior to start of study medication, except for participants who have been treated with interferon and in whom the ANC has fully recovered. Participants with neutropenia or thrombocytopenia in the last year, which resolved with splenectomy, may be considered for this study.
* Those who refuse to participate in the screening procedures or who are unable to participate in screening procedures or who are unable to comply with requirements of the protocol.
* Receiving other investigational products.
* Those in the opinion of the Investigator, who represent poor medical, psychological or psychiatric risks for whom participation in an investigational trial would be unwise.
* Those who are pregnant, breastfeeding or planning to become pregnant during the study period.
* Metallic objects in his/her body, such as artificial joints, inner ear (cochlear) implants, brain aneurysm clips, pacemakers, and metallic foreign bodies in the eye or other body areas.
* History of malignancy.
* Participants with claustrophobia.
* History of alcohol or drug abuse.
* Participants who are, in the opinion of the Investigator, excessively obese.

Ages: 18 Years to 36 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2002-12; Study Completion 2004-10

PRIMARY OUTCOMES:
To determine whether deferiprone exhibits superior efficacy in removing excess iron from the heart compared to that of deferoxamine, as reflected by MRI T2* assessments in the heart in participants treated with either chelator

SECONDARY OUTCOMES:
To evaluate the relative efficacy of deferiprone with respect to that of deferoxamine as assessed by serum ferritin concentration and liver iron concentration (LIC)

CONTACTS AND LOCATIONS:
Overall Officials: Renzo Galanello, M.D., Principal Investigator — Ospedale Regionale Microcitemie, Cagliari, Italy; Antonio Piga, M.D., Principal Investigator — Dipartimento di Scienze Pediatriche e Dell'Adolescenza, University of Turin, Turin, Italy; Markissia Karagiorga, M.D., Principal Investigator — Aghia Sophia Children's Hospital, Athens, Greece; Vassilis Ladis, M.D., Principal Investigator — 1st Department of Pediatrics, Athens University, Aghia Sophia Children's Hospital, Athens, Greece
Locations (4):
- Greece (2):
  - 1st Department of Pediatrics, Athens University, Aghia Sophia Children's Hospital, Athens
  - Aghia Sophia Children's Hospital, Athens
- Italy (2):
  - Ospedale Regionale Microcitemie, Dipartimento di Scienze, Cagliari, Sardinia
  - Dipartimento di Scienze e Dell' Adolescenza, University of Turin, Turin